CLINICAL TRIAL: NCT04843371
Title: Photoplethysmography (PPG) to Predict Ejection Fraction and Other Echographic Data in the General Population
Brief Title: PPG to Predict Ejection Fraction and Other Echographic Data in the General Population
Status: Recruiting | Type: Observational
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-441
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Valvular Heart Disease; Pericardial Disease; Cardiomyopathies
Keywords: Structural heart disease; Photoplethysmography; Ejection Fraction
MeSH Terms: conditions — Heart Valve Diseases; Cardiomyopathies | interventions — Photoplethysmography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Group: All patients undergoing an echocardiogram at Tulane Medical Center may be asked to participate in the study. Doctors, including PI and co-PI, will identify eligible patients from their clinic using their clinical knowledge and expertise and the patients' medical history and records. They will provide patients with information regarding the study and if interested, patients will be consented prior to their scheduled echocardiogram.
  Interventions: Diagnostic Test: Photoplethysmography

INTERVENTIONS:
Diagnostic Test: Photoplethysmography — Photoplethysmography (PPG) is a non-invasive technique that can detect volumetric changes in the peripheral blood. It only requires skin contact and relies on light absorption. PPG is a good indicator of the cardiovascular dynamics in the human body. PPG has been incorporated into various new smartphones and wearable devices such as, smartwatches and fitness wristbands making it readily available to all consumers. This sensor can record biometrics such as, heart rate, blood pressure, oxygen saturation, etc.

SUMMARY:
The investigators are aiming to investigate the association between ejection fraction (EF) determined by echocardiography and signals obtained from Photoplethysmography (PPG) in the general population. The investigators are also aiming to investigate the association between blood pressure and signals obtained from PPG in the general population.

Finally, the investigators are also aiming to investigate the association between signals obtained from PPG in the general population to cardioechographic findings such as, valvular heart disease, structural heart diseases, cardiomyopathies, pericardial disease etc.

DETAILED DESCRIPTION:
The investigators are proposing a cross-sectional cohort study, where any individual, 18 years old or older, scheduled for an echocardiography at Tulane University's outpatient cardiology clinic can be included. After consenting participants, information on their demographics, personal health habits, medications, and medical history will be collected via reviewing, their electronic medical health records. All participants will undergo an echocardiography as part of their routine medical care by their treating physician. Important echocardiographic findings will be noted such as, EF, valvular heart disease, pericardial disease, cardiomyopathies and structural heart disease. Additionally, PPG recordings will be collected simultaneously while performing echography using the Biostrap wristband.

The investigators will analyze the association between each echographic imaging feature, and the PPG waveform obtained. PPG waveform features will be used to develop a predictive model capable of calculating an estimate of ventricular ejection fraction without echocardiography. All echocardiograms will be performed by experienced operators at Tulane Medical Center facilities. The study will occur at a single study site Tulane Medical Center and clinics, with appropriate facilities and equipment to conduct the study accurately and safely.

An experienced echocardiogram technician or cardiology fellow will collect the PPG recordings using the Biostrap application. De-identified echocardiogram reports, including information on LVEF will be matched with the participant's pulse report.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged18 years or older.
* Patients scheduled to undergo an echocardiogram at Tulane Medical Center.

Exclusion Criteria:

* Participants under 18 years of age.
* Participants with cognitive impairments.
* Participants with a physical inability to wear the Biostrap during the echocardiogram.
* Individuals who cannot read, speak, and/or understand English.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing an echocardiogram at Tulane Medical Center may be asked to participate in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Association between obtained PPG waveforms and recorded ejection (EF) fractions. | Day 1
  Patients who will undergo echocardiogram will wear the biostrap watch and then the PPG waveform will be obtained. Then, the ejection fraction will be collected from the echocardiogram report. Then, the Artificial Intelligence (AI) staff member will do a predictive model to try and estimate the EF based on the PPG waveform.

SECONDARY OUTCOMES:
Association between blood pressure and PPG waveforms | Day1
  The investigators will record the blood pressure of the patient twice during their visit. Then, the Artificial Intelligence (AI) staff member will do a predictive model to try and estimate the blood pressure based on the PPG waveform.

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Marrouche, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane University Medical Center, New Orleans, Louisiana, United States

REFERENCES:
- [Background] McDonagh TA, McDonald K, Maisel AS. Screening for asymptomatic left ventricular dysfunction using B-type natriuretic Peptide. Congest Heart Fail. 2008 Jul-Aug;14(4 Suppl 1):5-8. doi: 10.1111/j.1751-7133.2008.tb00002.x. PMID 18772638
- [Background] Dargie HJ. Effect of carvedilol on outcome after myocardial infarction in patients with left-ventricular dysfunction: the CAPRICORN randomised trial. Lancet. 2001 May 5;357(9266):1385-90. doi: 10.1016/s0140-6736(00)04560-8. PMID 11356434
- [Background] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliott PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ; ESC Scientific Document Group. 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC). Eur Heart J. 2015 Nov 1;36(41):2793-2867. doi: 10.1093/eurheartj/ehv316. Epub 2015 Aug 29. No abstract available. PMID 26320108
- [Background] Betti I, Castelli G, Barchielli A, Beligni C, Boscherini V, De Luca L, Messeri G, Gheorghiade M, Maisel A, Zuppiroli A. The role of N-terminal PRO-brain natriuretic peptide and echocardiography for screening asymptomatic left ventricular dysfunction in a population at high risk for heart failure. The PROBE-HF study. J Card Fail. 2009 Jun;15(5):377-84. doi: 10.1016/j.cardfail.2008.12.002. Epub 2009 Jan 21. PMID 19477397
- [Background] Redfield MM, Rodeheffer RJ, Jacobsen SJ, Mahoney DW, Bailey KR, Burnett JC Jr. Plasma brain natriuretic peptide to detect preclinical ventricular systolic or diastolic dysfunction: a community-based study. Circulation. 2004 Jun 29;109(25):3176-81. doi: 10.1161/01.CIR.0000130845.38133.8F. Epub 2004 Jun 7. PMID 15184280
- [Background] Blanie A, Soued M, Benhamou D, Mazoit JX, Duranteau J. A Comparison of Photoplethysmography Versus Esophageal Doppler for the Assessment of Cardiac Index During Major Noncardiac Surgery. Anesth Analg. 2016 Feb;122(2):430-6. doi: 10.1213/ANE.0000000000001113. PMID 26649910
- [Background] Chan GS, Middleton PM, Celler BG, Wang L, Lovell NH. Automatic detection of left ventricular ejection time from a finger photoplethysmographic pulse oximetry waveform: comparison with Doppler aortic measurement. Physiol Meas. 2007 Apr;28(4):439-52. doi: 10.1088/0967-3334/28/4/009. Epub 2007 Mar 20. PMID 17395998
- [Background] Middleton PM, Chan GS, O'Lone E, Steel E, Carroll R, Celler BG, Lovell NH. Changes in left ventricular ejection time and pulse transit time derived from finger photoplethysmogram and electrocardiogram during moderate haemorrhage. Clin Physiol Funct Imaging. 2009 May;29(3):163-9. doi: 10.1111/j.1475-097X.2008.00843.x. Epub 2009 Jan 22. PMID 19170720
- [Background] Nachman D, Gepner Y, Goldstein N, Kabakov E, Ishay AB, Littman R, Azmon Y, Jaffe E, Eisenkraft A. Comparing blood pressure measurements between a photoplethysmography-based and a standard cuff-based manometry device. Sci Rep. 2020 Sep 30;10(1):16116. doi: 10.1038/s41598-020-73172-3. PMID 32999400